CLINICAL TRIAL: NCT05508971
Title: Treatment of Obstructive Sleep Apnea With Personalized Surgery in Children With Down Syndrome (TOPS-DS)
Acronym: TOPS-DS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); University of Michigan (Other); University of Texas (Other); Eastern Virginia Medical School (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Texas Children's (Unknown); Children's Hospital Colorado (Other)
Responsible Party: Principal Investigator, Derek Lam, MD, MPH, Associate Professor of Otolaryngology - Head and Neck Surgery, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00024746; 1R61HL165345 (NIH)
Record Dates: First submitted 2022-08-10; First posted 2022-08-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Obstructive Sleep Apnea; Down Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive; Down Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be recruited from pediatric otolaryngology clinics. The study will be introduced to caregivers of children with DS and a history of sleep disordered breathing/OSA who are referred for surgery and meet the study participation criteria noted. If current or recent PSG testing demonstrates OSA, they will be invited to participate.
  Randomization will be done. Patients will be randomized to either the personalized DISE-directed surgery or the standard AT after collection of baseline measures and pre-op PSG. Allocation will be made by using a computer-generated randomization scheme. Caregivers will be advised of the outcomes and risks of different surgical procedures included in DISE-directed surgery and informed consent will be obtained. All patients will be planned for overnight observation to monitor for safety and periop complications.
Who Masked: Outcomes Assessor
Masking Description: It is not practical or feasible to maintain blinding among the surgeons performing the procedures or the clinical staff caring for patients in the perioperative setting. Given this, it is unlikely that blinding could be maintained among parents or caregivers of patients, therefore there will be no attempt to blind caregivers to the treatment assignment. However, the sleep medicine collaborators who will be reviewing and scoring postoperative PSGs will be instructed not to review the medical record so as to ensure blinding to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug-Induced Sleep Endoscopy (Experimental): DISE will be performed at the time of surgery under the same sedation. The decision on specific surgical approach will be made at that time based on DISE findings. Prior to intubation, patients will be sedated with either a propofol infusion or a combination of ketamine and dexmedetomidine. Once adequate sedation is achieved, endoscopy will be performed using a flexible endoscope advanced through the nose. The nasal airway will be evaluated on both sides, then the endoscope will be advanced into the pharynx. The degree of obstruction is scored on a 3-point rating scale. Participants randomized to DISE-directed surgery will undergo one or more potential procedures in a single surgery. Caregivers will be consented for all possible procedures with the understanding that only those needed based on DISE will be performed. Importantly, these procedures are all established treatments with published outcomes data.
  Interventions: Procedure: DISE-Directed Surgery
- Adenotonsillectomy (Active Comparator): Adenotonsillar hypertrophy is the most common risk factor for OSA in children, and adenotonsillectomy (AT) is the first line treatment. An adenotonsillectomy is an operation to remove both the adenoids and tonsils.
  Interventions: Procedure: Adenotonsillectomy

INTERVENTIONS:
Procedure: DISE-Directed Surgery — Participants randomized to DISE-directed surgery will undergo one or more potential procedures in a single surgery (i.e. DISE and subsequent sleep surgery performed) concurrently under the same general anesthetic), depending on anatomic assessment.
  Arms: Drug-Induced Sleep Endoscopy
Procedure: Adenotonsillectomy — Tonsil and adenoid removal
  Other Names: AT
  Arms: Adenotonsillectomy

SUMMARY:
The overall objective of this randomized clinical trial is to test the effectiveness of a personalized approach to the surgical treatment of OSA in children with Down syndrome (DS).The estimated prevalence of obstructive sleep apnea (OSA) in children with DS ranges from 45-83%, compared to 1-6% in the general pediatric population. Untreated OSA in children has been associated with daytime sleepiness, cognitive or behavioral problems, and cardiovascular complications, all which are common in children with DS. Adenotonsillectomy (AT) is the first line treatment for OSA in children, however, most large studies of AT outcomes have excluded children with DS. Available evidence demonstrates that AT is far less effective in children with DS than in the general pediatric population, with 48 to 95% of children with DS having persistent OSA after AT. Medical treatments such as positive airway pressure (PAP) therapy are frequently inadequate or poorly tolerated in this population, so many children with DS and OSA remain untreated. Drug-induced sleep endoscopy (DISE) enables direct observation of the sites and patterns of obstruction during sedated sleep using a flexible endoscope passed through the nose into the pharynx. DISE was developed to guide surgical decisions in adult OSA, and in recent years has also been used to design personalized surgical interventions in children. Using this DISE Rating Scale, the investigators have demonstrated that children with DS are more prone to tongue base and supraglottic obstruction than non-DS children, suggesting the need for more personalized surgical treatments that are tailored to the common sources of obstruction in this population. Several small case series demonstrate that DISE-directed surgery can be effective in treating OSA in children with DS. However, because there have been few prospective studies and no randomized trials comparing different treatment options in this population, there remains uncertainty about whether such a personalized approach leads to superior outcomes compared to the first line AT.

It is the investigators' hypothesis that personalized DISE-directed surgery that uses existing procedures to address specific fixed and dynamic anatomic features causing obstruction in each child with DS will be superior to the current first line approach of AT. This novel approach may improve OSA outcomes and reduce the burden of unnecessary AT or secondary surgery for persistent OSA after an ineffective AT.

DETAILED DESCRIPTION:
The overall objective of this randomized clinical trial is to test the effectiveness of a novel personalized approach to the surgical treatment of OSA in children with Down syndrome (DS). DS is a common disorder, affecting 1 in 691 births. The estimated prevalence of obstructive sleep apnea (OSA) in children with DS ranges from 45-83%, compared to 1-6% in the general pediatric population. Untreated OSA in children has been associated with daytime sleepiness, cognitive and behavioral problems, and cardiovascular complications, all of which are common in children with DS. Adenotonsillectomy (AT) is the first line treatment for OSA in children, however, most large studies of AT outcomes have excluded children with DS. Available evidence demonstrates that AT is far less effective in children with DS than in the general pediatric population, with 48 to 95% of children with DS having persistent OSA after AT. Medical treatments such as positive airway pressure (PAP) therapy are frequently inadequate or poorly tolerated in this population, so many children with DS and OSA remain untreated.

Pharyngeal hypotonia, unfavorable craniofacial anatomy, and adiposity are commonly cited risk factors for OSA and failure of AT in children with DS, however, there have been few attempts to characterize the pharyngeal anatomy or mechanisms of obstruction in this population. Drug-induced sleep endoscopy (DISE) enables direct observation of the sites and patterns of pharyngeal obstruction during sedated sleep using a flexible endoscope passed through the nose into the pharynx. DISE was developed to guide surgical decisions in adult OSA, and in recent years has also been used to design personalized surgical interventions in children. To help standardize DISE assessments, the investigators previously developed and validated the DISE Rating Scale in children based on ordinal ratings of maximal airway obstruction (none, partial, complete) at six anatomic sites from the nose to the larynx. Using this DISE Rating Scale, the investigators have demonstrated that children with DS are more prone to tongue base and supraglottic obstruction than non-DS children, suggesting the need for more personalized surgical treatments that are tailored to the common sources of obstruction in this population. Several small case series demonstrate that DISE-directed surgery can be effective in treating OSA in children with DS. However, because there have been few prospective studies and no randomized trials comparing different treatment options in this population, there remains uncertainty about whether such a personalized approach leads to superior outcomes compared to the first line AT.

It is the investigators' central hypothesis that a personalized DISE-directed surgical approach that uses existing procedures to address the specific fixed and dynamic anatomic features causing obstruction in each child with DS will be superior to the currently recommended first line approach of AT. This novel approach may improve OSA outcomes and reduce the burden of unnecessary AT or secondary surgery for persistent OSA after an ineffective AT.

To test this hypothesis, the investigators propose to study children with DS and OSA ages 2-17 years with the following specific aims:

Aim 1: Compare the physiological outcomes of DISE-directed surgery vs AT in children with DS and OSA.

Hypothesis 1: DISE-directed surgery will result in a greater improvement in the obstructive apnea-hypopnea index compared to the standard AT intervention (effect size ≥ 0.36) after 6 months.

Aim 2: Compare the clinical outcomes of DISE-directed surgery vs AT in children with DS and OSA.

Hypothesis 2: DISE-directed surgery will result in a clinically significantly greater improvement (≥ 9 point improvement) in OSA-specific quality of life (OSA-18) compared to the standard AT intervention after 6 months. Secondarily, the investigators will test other clinical outcomes such as executive function (BRIEF2).

The investigators propose a randomized single-blind comparative effectiveness trial of AT vs DISE-directed sleep surgery for the treatment of OSA in children with DS (Figure 4). The investigators' primary hypothesis is that a personalized surgical intervention based on DISE findings will be more effective in treating OSA in children with DS than the standard AT. The first aim will compare the change in the obstructive apnea-hypopnea index (oAHI) between these treatment arms, and the second aim will compare the change in subjective measures of sleep apnea related quality of life (OSA-18) and executive function (BRIEF2). Outcomes will be assessed 6 months after surgery. The trial will be conducted at seven sites: Oregon Health and Science University, Cincinnati Children's Hospital and Medical Center, University of Michigan, University of Texas-Southwestern, Eastern Virginia Medical School, Texas Children's, and Children's Hospital Colorado.

ELIGIBILITY:
Requirements to participate in study:

Child has a diagnosis of Down syndrome (Trisomy 21). Child has a diagnosis of moderate to severe OSA diagnosed by PSG (oAHI ≥ 5). Child age is 2.00 to 17.99 years of age. Caregiver can provide signed and dated consent and is 18 years of age or older at the time of consent.

Caregiver can speak, read, and write in English or Spanish. Caregiver is primary caretaker of the child. Child is not expecting their own child. Child is eligible for surgical treatment

Cannot participate in study if:

Child has history of previous tonsillectomy, tonsillotomy, or partial tonsillectomy.

Child has any contraindication to surgery (e.g. bleeding disorders). Child has significant cardiopulmonary comorbidity besides OSA requiring supplemental oxygen, subglottic or tracheal stenosis, tracheostomy dependence.

Caregiver is unwilling or unable to comply with study procedures. Child is or plans to have their own child.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 303 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Polysomnography Measures: oAHI at 6 months | 6 month follow up sleep study (after surgery)
  Objective results from sleep studies (polysomnography): Obstructive Apnea-Hypopnea Index (oAHI): 6 months follow up sleep study difference from baseline sleep study
Change from Baseline Polysomnography Measures: AHI at 6 months | 6 month follow up sleep study (after surgery)
  Objective results from sleep studies (polysomnography): Total Apnea-Hypopnea Index: 6 months follow up sleep study difference from baseline sleep study
Change from Baseline Polysomnography Measures: REM AHI at 6 months | 6 month follow up sleep study (after surgery)
  Objective results from sleep studies (polysomnography): REM Apnea-Hypopnea Index REM AHI: 6 months follow up sleep study difference from baseline sleep study
Change from Baseline Polysomnography Measures: min SpO2 at 6 months | 6 month follow up sleep study (after surgery)
  Objective results from sleep studies (polysomnography): Minimum Oxygen Saturation (Min SpO2): 6 months follow up sleep study difference from baseline sleep study
Change from Baseline Polysomnography Measures: desat index at 6 months | 6 month follow up sleep study (after surgery)
  Oxyhemoglobin desaturation ≥ 3% Index: 6 months follow up sleep study difference from baseline sleep study
Change from Baseline Polysomnography Measures: % Total Sleep Time with ETCO2 > 50 mmHg at 6 months | 6 month follow up sleep study (after surgery)
  % Total Sleep Time with ETCO2 > 50 mmHg: 6 months follow up sleep study difference from baseline sleep study
Change from Baseline Polysomnography Measures: Max End Tidal CO2 (ETCO2) at 6 months | 6 month follow up sleep study (after surgery)
  Max End Tidal CO2 (ETCO2): 6 months follow up sleep study difference from baseline sleep study

SECONDARY OUTCOMES:
Change in Obstructive Sleep Apnea (OSA)-18 Questionnaire score | 6 month follow up
  Disease specific quality of life measure: 18 questions, scores range from 18-126; higher scores means higher disease burden
Change in Generic PedsQL (Pediatric Quality of Life) Questionnaire score | 6 month follow up
  Generic quality of life measure: an age specific questionnaire with 23 questions (scores range from 0-100); higher scores indicate better quality of life.
Change in Generic PedsQL (Pediatric Quality of Life) Questionnaire answers | 6 month follow up
  Quality of life: questionnaire results by individual question. Adjusted scores range from 0-100; higher scores indicate better quality of life.
Total Drug induced sleep endoscopy (DISE) score | At time of surgery
  Subjective ratings of degree of obstruction at 6 levels of the upper airway, done by surgeon. Scores range from 0 to 12. Higher scores means more breathing obstruction, or more disease burden.
Adverse Events | 24 hour period after surgery
  Did any adverse events occur in the post-operative time frame? This is a yes/no question, looking at the following outcomes: dehydration and poor oral intake due to post-operative pain, post-tonsillectomy hemorrhage, and respiratory compromise.
  respiratory compromise.
Change in Feeding and Swallowing Impact Survey (FSIS) Questionnaire Answers | 6 month follow up
  Dysphagia specific quality of life measure: 18 questions, scores range from 18-90; higher scores means higher disease burden.

CONTACTS AND LOCATIONS:
Overall Officials: Derek Lam, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (7):
- United States (7):
  - Colorado Children's Hospital, Aurora, Colorado
  - University of Michigan, Ann Arbor, Michigan
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - EVMS Medical School, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No
IPD will not be made available to researchers who are not primary researchers on this study.